CLINICAL TRIAL: NCT05598151
Title: A Phase I, Open-Label, Multicenter, Dose Escalation and Expansion Study of HM97662 as a Single Agent in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation and Expansion Study of HM97662 in Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-EZHI-101
Record Dates: First submitted 2022-09-05; First posted 2022-10-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HM97662 (Experimental): Tablet, oral administration, once daily (QD), continuous dosing
  Interventions: Drug: HM97662

INTERVENTIONS:
Drug: HM97662 — To evaluate the safety, tolerability, preliminary anti-tumor efficacy, PK and PD of HM97662 in solid tumors

SUMMARY:
This is a Phase1 study to assess the safety, PK, PD and efficacy of HM97662, EZH1/2 dual inhibitor, in solid tumors. The study is comprised of Dose-Escalation Part followed by randomized Dose-Ranging Part and Dose-Expansion Part. Dose-Escalation Part is planned with a 3+3 Dose-Escalation design and is to establish the MTD or RD for randomized Dose-Ranging Part. Dose-Ranging Part is designed mainly to further evaluate safety and preliminary efficacy of HM97662 monotherapy in subjects with specific genomic alterations to more precisely determine the potential RP2D that are to be tested in a Dose-Expansion Part. Dose-Expansion Part is designed to assess the potential efficacy of HM97662 monotherapy when administered at the RP2D to subjects in indication-specific expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed advanced or metastatic solid tumor who have failed/are intolerant to standard therapy.
* Patients for dose-escalation part must have evaluable or measurable disease at baseline and the patients for randomized dose-ranging and dose-expansion part must have at least one measurable lesion at baseline by CT or MRI per Response Evaluation Criteria in Solid Tumor (RECIST v1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥ 3 months before starting HM97662.
* Adequate renal function.
* Adequate hematologic function.
* Adequate liver function.
* Males or females aged ≥ 18 years (or country's legal age of majority if the legal age was > 18 years) at the time of informed consent.
* For Dose-Ranging Part, documentation of an alteration in at least one of the genes of the SWI/SNF complex in tumor tissue (archival or newly obtained).

Exclusion Criteria:

* Prior exposure to valemetostat or other EZH1/2 dual inhibitor.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms.
* Patients currently taking medications that are known strong CYP3A inhibitors and strong or moderate CYP3A inducers.
* Any prior treatment-related (i.e. chemotherapy, immunotherapy, radiotherapy) clinically significant toxicities that have not resolved to Grade ≤ 1 per CTCAE version 5.0 or prior treatment-related toxicities that are clinically unstable and clinically significant at time of enrollment.
* Major surgery within 4 weeks before the first dose of study drug treatment in Cycle 1.
* Females who are pregnant or breastfeeding.
* Patients who have undergone an organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of DLTs | Days 1-28 of Cycle 1 (DLT assessment period) in Dose-Escalation Part
Incidence, nature, and severity of adverse events and laboratory abnormalities graded per NCI CTCAE v5.0 | until Safety Follow-up, 30 days after the last dose of study drug or until initiation of another anti-cancer therapy, whichever occurs first

SECONDARY OUTCOMES:
Area under the concentration-time curve (AUC) | until Cycle 4 Day1 (each cycle is 28 days)
The maximum plasma concentration (Cmax) | until Cycle 4 Day1 (each cycle is 28 days)
Trough plasma concentration (Ctrough) | until Cycle 4 Day1 (each cycle is 28 days)
Time to reach Cmax (Tmax) | until Cycle 4 Day1 (each cycle is 28 days)
Terminal Half-life (T1/2) | until Cycle 4 Day1 (each cycle is 28 days)
Apparent clearance (CL/F) | until Cycle 4 Day1 (each cycle is 28 days)
Apparent volume of distribution (Vd/F) | until Cycle 4 Day1 (each cycle is 28 days)
Objective response | Day 1 of Cycles 3, 5, 7 (each cycle is 28 days) and further (every 8 weeks) until disease progression (assessed up to 5 years)

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (4):
  - Cancer Research SA, Adelaide
  - Grampians Health, Ballarat
  - Monash Medical Centre, Clayton
  - Peninsula and Southeast Oncology, Frankston
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul